CLINICAL TRIAL: NCT01882959
Title: Radiofrequency Denervation for Reducing Chronic Pain: a Meta-analysis
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: RF_META
Record Dates: First submitted 2013-06-18; First posted 2013-06-21 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Neck Pain; Chronic Low Back Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Placebo
- Intervention: Radiofrequncy Denervation
  Interventions: Other: Radiofrequncy Denervation

INTERVENTIONS:
Other: Radiofrequncy Denervation
  Groups: Intervention

SUMMARY:
The meta-analysis of data obtained from randomized controlled trial on effectiveness of radiofrequency denervation on reducing chronic neck and low back pain.

ELIGIBILITY:
Inclusion Criteria:

* RCTs with pain VAS as outcome

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with chronic neck or low back pain.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 2013-01; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analogue Scale | 4 months